CLINICAL TRIAL: NCT06610331
Title: EVALUATION OF THE EFFECT OF POLYVINYLPYROLIDONE AND SODIUM HYALURONATE GEL ON PALATINAL WOUND HEALING: A RANDOMIZED CONTROLLED CLINICAL STUDY
Brief Title: EVALUATION OF THE EFFECT OF POLYVINYLPYROLIDONE AND SODIUM HYALURONATE GEL ON PALATINAL WOUND HEALING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, nuray Ercan, ASSISTANT PROFESSOR, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BAIBU-SBF-NE-01
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Palatal Wound
Keywords: WOUND HEALİNG; sodium hyaluronate; Polyvinylpyrrolidone; Free gingival graft; PALATAL

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control Group - Free Gingival Graft (Sham Comparator)
  Interventions: Procedure: FREE GİNGİVAL GRAFT
- Test Group - Free Gingival Graft + polyvinylpyrrolidone sodium hyaluronate gel (Experimental)
  Interventions: Procedure: FREE GİNGİVAL GRAFT; Device: polyvinylpyrrolidone sodium hyaluronate gel

INTERVENTIONS:
Procedure: FREE GİNGİVAL GRAFT — Free Gingival Graft removal from the palate donor area for the treatment of gingival recession
Device: polyvinylpyrrolidone sodium hyaluronate gel — Patients are told to gargle with a mouthwash containing polyvinyl pyrrolidone sodium hyaluronate twice a day for 2 weeks. 15 ml (1 tablespoon) of mouthwash containing polyvinyl pyrrolidone sodium hyaluronate is poured into a glass and approximately 40 ml (3 tablespoons) of water is added and mixed well, then it is shaken for at least 1 minute, making contact with the entire mouth.
  Arms: Test Group - Free Gingival Graft + polyvinylpyrrolidone sodium hyaluronate gel

SUMMARY:
The aim of this clinical study was to evaluate the effect of polyvinylpyrrolidone sodium hyaluronate gel on palatal wound healing, pain, and bleeding after free gingival graft surgery. This study included 32 systemically healthy patients who required free gingival graft surgery. After the operation, the test group received polyvinylpyrrolidone sodium hyaluronate gel in addition to chlorhexidine gluconate mouthwash, whereas the control group received only chlorhexidine gluconate mouthwash. VAS scale was used to evaluate palatal pain, burning, and chewing discomfort, WHI was used to evaluate wound healing, and H2O2 foaming test was used to evaluate epithelialization. VAS and bleeding values were recorded on postoperative day 1; VAS, WHI, H2O2, and bleeding values on postoperative days 3, 7, and 14; and WHI, H2O2, and bleeding values on postoperative day 28.

ELIGIBILITY:
Inclusion Criteria:

* Able to adapt to the study, not having a physical or psychological condition that would prevent surgical procedure under local anesthesia, and being able to follow the planned operation and control sessions
* Patients who consciously accept and sign the detailed informed consent form regarding the study that will be explained to them verbally
* Insufficiently attached gingiva on the mandibular or maxillary vestibular teeth and implant surfaces

Exclusion Criteria:

* Presence of infection and inflammation in the recipient and donor area
* Presence of systemic disease
* Women who are pregnant, suspected of being pregnant or breastfeeding
* Smoking
* Orofacial neurological symptoms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Epithelialization | 28 days
  Epithelialization of the palatal region was performed by applying 3% hydrogen peroxide to the wound area with the help of an injector, and the areas showing foaming (H2O2 bubbling) in the total surface area of the wound area were calculated as a percentage and recorded, providing information about epithelialization.

SECONDARY OUTCOMES:
wound healing | 28 days
  Palatal wound healing was assessed using the Wound Healing Index (WHI) as described by Landry et al. (1985)

CONTACTS AND LOCATIONS:
Locations (1):
- Bolu Abant Izzet Baysal University Faculty of Dentistry Department of Periodontology, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bulut T, Ercan N. The effect of Polyvinylpyrrolidone-Sodium hyaluronate gel on palatal wound healing: a randomized controlled clinical trial. BMC Oral Health. 2025 Aug 8;25(1):1305. doi: 10.1186/s12903-025-06677-w. PMID 40781616